CLINICAL TRIAL: NCT04614558
Title: A Single Arm, Multicenter, Phase II, Open-Label Trial to Evaluate Efficacy of Isatuximab in Patients With Monoclonal Gammopathy of Renal Significance
Brief Title: Isatuximab in Patients With Monoclonal Gammopathy of Renal Significance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Divaya Bhutani, Assistant Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT0761
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Monoclonal Gammopathy
MeSH Terms: conditions — Paraproteinemias | interventions — isatuximab

STUDY DESIGN:
Intervention Model Description: The study will be a single arm, prospective, multi-center, phase II, open- label study including 27 subjects in total. The study will consist of a screening phase, treatment phase, post-treatment observation phase and follow-up phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isatuximab for MGRS (Experimental): Subjects will receive Isatuximab for 6 months and will be followed for an additional one year post therapy for outcome follow-up.
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — Isatuximab in IV form (10mg/kg q weekly x 4 doses followed by 10mg/kg q 2 weeks) for a total of 6 month duration. Doses should be initiated at 175 mg/hour up to a maximum of 400 mg/hour.
  Isatuximab (SAR) is monoclonal antibody (mAb).
  Other Names: Sarclisa

SUMMARY:
The purpose of this study is to see whether Isatuximab can help improve kidney function of participants with MGRS. Isatuximab is approved by the Food and Drug Administration (FDA) for the treatment of adult patients with multiple myeloma, but it is not approved by the FDA to treat MGRS. This means that the use of isatuximab in this study is considered 'investigational'.

DETAILED DESCRIPTION:
Monoclonal gammopathy is a common disorder but only a small fraction of patients with monoclonal gammopathy of undetermined significance (MGUS) develop renal disease and the reason for abnormal deposition of immunoglobulin in renal parenchyma remains unclear in these disorders. The proposed research will be conducted as a part of clinical trial which intends to prospectively evaluate the effect of anti-plasma cell therapy on renal outcomes in patients with monoclonal gammopathy of renal significance (MGRS). The study specifically intends to sequence the immunoglobulin heavy and light chain genes to determine any abnormalities that could lead to production of a misfolded immunoglobulin thus leading to deposition in renal parenchyma.

ELIGIBILITY:
Inclusion Criteria:

1. Renal biopsy proven diagnosis of an MGRS disorder including the following:

   1. Proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMID)
   2. C3 glomerulopathy associated with monoclonal gammopathy
   3. Non-Amyloid Fibrillary Glomerulonephritis
   4. Light chain Proximal Tubulopathy
   5. Immunotactoid Glomerulopathy

   A concurrent diagnosis of Monoclonal gammopathy (with +ve Serum and/or Urine protein electrophoresis or Bone marrow biopsy) is required in patients with C3 glomerulopathy but not for other disorders. Patients with concurrent MGUS, non-high risk smoldering myeloma are eligible for enrollment.
2. Measurable Proteinuria ≥1gram over 24 hours.
3. Prior Therapy: Newly diagnosed as well as patients with previous therapy but persistent renal dysfunction and persistent proteinuria ≥1gram over 24 hours are eligible for enrollment. Patients who received a prior cluster of differentiation 38 (CD38) antibody therapy are not eligible for study. In patients who have received prior therapy a wash out period of 12 weeks for chemotherapy based therapies and 24 weeks for Rituximab based therapies is required between completion of prior therapy and cycle 1 Day1 of study therapy.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Life expectancy of greater than 6 months
7. Participants must have normal organ and marrow function as defined below:

Leukocytes ≥3,000/microliters (mcL)

1. absolute neutrophil count ≥1,500/mcL
2. platelets ≥100,000/mcL
3. total bilirubin within normal institutional limits
4. Aspartate aminotransferase (AST) (SGOT)/alanine transaminase (ALT)(SGPT) ≤2.5 × institutional upper limit of normal
5. Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2.

Exclusion Criteria:

1. Participants who have had chemotherapy based therapy within 12 weeks or Rituximab based therapy within prior 24 weeks prior to starting the cycle 1 Day 1 of trial therapy
2. Participants who are receiving any other investigational agents concurrently.
3. History of severe allergic reactions or anaphylaxis attributed to compounds of similar chemical or biologic composition to Isatuximab.
4. Diagnosis of Multiple Myeloma or High risk smoldering Multiple Myeloma or a B cell lymphoma meeting criteria for therapy.
5. Renal Biopsy showing the coexistence of other significant diagnosis e.g. diabetic nephropathy.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant and Lactating women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Isatuximab.
8. HIV-positive Participants are ineligible because of increased risk of lethal infections when treated with immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Renal Response Rate | Up to 6 months
  Renal response defined as a decrease in 24-hour proteinuria by >50% at any point post therapy.

SECONDARY OUTCOMES:
Number of Adverse Events | Up to 12 months
  The number of adverse events recorded for participants using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Percentage of Participants with Immunoglobulin Gene Mutations | Baseline, up to 4 weeks prior to treatment
  The percentage of participants with immunoglobulin gene mutations as determined by next generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Divaya Bhutani, MD, Principal Investigator — Assistant Professor of Medicine at the Columbia University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Renal Associates Clinic, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No